CLINICAL TRIAL: NCT01303926
Title: Induction Pemetrexed and Cisplatin Followed by Pemetrexed as Maintenance vs Carboplatin-paclitaxel and Bevacizumab Followed by Bevacizumab as Maintenance:Multicenter Randomized Phase III Study in Patients With Advanced Non-Squamous Non Small-cell Lung Cancer: a Quality of Life Oriented Phase III Trial of the GOIM
Brief Title: Quality of Life Comparison in Advanced Non-squamous Non Small Cell Lung Cancer
Acronym: ERACLE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gruppo Oncologico Italia Meridionale (Other)
Responsible Party: Principal Investigator, Giuseppe Colucci MD, President, Gruppo Oncologico Italia Meridionale
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Goim 2903; 2009-015807-19 (EudraCT Number)
Record Dates: First submitted 2011-01-13; First posted 2011-02-25 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-04

CONDITIONS: Non-squamous Nonsmall Cell Neoplasm of Lung
Keywords: QoL; EQ5D score; cisplatin pemetrexed; carboplatin paclitaxel bevacizumab; maintenance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cisplatin and Pemetrexed (Active Comparator)
  Interventions: Drug: cisplatin pemetrexed
- Carboplatin paclitaxel bevacizumab (Active Comparator)
  Interventions: Drug: carboplatin paclitaxel bevacizumab

INTERVENTIONS:
Drug: cisplatin pemetrexed — Cisplatin 75 mg / m2 d1 with Pemetrexed 500 mg / m2 d1 every 3 weeks for 6 cycles followed (in responding or stable patients) by Pemetrexed 500 mg / m2 every 3 weeks, until progression or unacceptable toxicity
  Arms: Cisplatin and Pemetrexed
Drug: carboplatin paclitaxel bevacizumab — Carboplatin AUC 6 d1 plus Paclitaxel 200 mg/m2 d1 and Bevacizumab 15 mg/kg every 3 weeks for 6 cycles followed in stable or responding patients by Bevacizumab 15 mg/kg every 3 weeks, until progression or unacceptable toxicity
  Arms: Carboplatin paclitaxel bevacizumab

SUMMARY:
Cisplatin and pemetrexed combination or carboplatin, paclitaxel and bevacizumab are now considered as standard treatment in non-squamous cell lung carcinoma (NSCLC). Both main registrative trials are considered positive because they reached their objectives, but within them, the Quality of Life (QoL) of patients was not detailed neither has represented as primary objective of the studies. It is considered that, together with enhancements that are added to the knowledge of the biology of NSCLC, QoL may influence the therapeutic choice if one of the associations show to be better tolerated by the patient and favours an amelioration of his QoL.

DETAILED DESCRIPTION:
The study aims primarily to verify the null hypothesis that between the two schemes under consideration there is no minimal interesting difference (MID) (i.e. a difference of clinical interest) after initial 3 months of maintenance.EuroQ5D (EQ5D) questionnaire total score and EQ5D visual analog scale (VAS)are validated and very simple to be administered.The statistical hypothesis tests described above are performed with t-test for unpaired data (or equivalent non-parametric, pending verification of normality of distribution by Shapiro-Wilk test), with alpha error = 0.05 (2-sided). It is assumed that:

1. about 20% of randomized patients experienced a progression of disease before the time of evaluation of the primary endpoint, and that
2. this eventuality was not significantly different between the two treatments. The total sample to be enrolled for this study will then be increased to 118 patients [(49 +49) +20%)]

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent(as approved by the local Ethical Committee)
* Histological type consisting mainly of non-squamous histology defined preferably with stage IV metastatic disease or stage IIIB in the presence of supraclavicular lymph nodes according to the parameters of TNM 7th Ed, not amenable to curative therapy
* ECOG PS 0-1
* Adequate bone marrow reserve
* Adequate hepatic, coagulative and renal function

Exclusion Criteria:

* Mixed NSCLC tumors or mixed adenosquamous carcinomas with a predominant squamous component histotype (NSCLC and SCLC) or adenosquamous forms, with predominant squamous component
* History of gross hemoptysis <3 months prior to enrollment or history or evidence of inherited bleeding diathesis or coagulopathy with the risk of bleeding.
* Tumors invading or abutting major blood vessels (based on radiologist assessment)
* Evidence of brain metastases not previously treated with RT (or any loco-regional treatment)
* Prior neoadjuvant or adjuvant chemotherapy within six months prior to study enrollment
* Previous radiotherapy in the last month before study entry (except for radiotherapy to symptomatic bone sites at risk and not covered in the premises of measurable disease and assessable)
* A major surgery (including open biopsy) in the month preceding study enrollment or anticipation of a major surgery during the study
* Unable or unwilling to take folic acid or vitamin B12 supplementation
* Unable or unwilling to take corticosteroids
* History of gastrointestinal fistula, perforation, or abscess, inflammatory bowel disease, or diverticulitis
* Clinically significant third-space fluid collections, for example, ascites or pleural effusions that cannot be controlled by drainage or other procedures prior to study entry
* Need for taking or have recently taken (within 10 days of enrollment) aspirin (>325 mg/d), clopidogrel at doses >75 mg/d, dipyramidole, ticlopidine, or cilostazol. Patients are also excluded if they cannot hold nonsteroidal anti-inflammatory agents, other than prophylactic therapy with low-dose aspirin, for a 5-day period during each cycle (8-day period for long-acting agents, such as piroxicam)
* Need for taking or have recently taken (within 10 days of enrollment) fulldose oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes. Prophylactic use of anticoagulants is allowed; international normalized ratio (INR) should be <1.5 at study enrollment
* History of thrombotic disorders within the last 6 months prior to entry History of hypertension, unless hypertension is well controlled study entry (≤150/90 mm Hg) and the patient is on a stable regimen of antihypertensive therapy. Patients should not have any prior history of hypertensive crisis or hypertensive encephalopathy
* Serious cardiac condition, such as myocardial infarction within 6 months, angina, or heart disease, as defined by the New York Heart Association Class III or IV
* Serious concomitant systemic disorder (for example, active infection including human immunodeficiency virus) that, in the opinion of the investigator, would compromise the patient's ability to adhere to the protocol
* Receiving concurrent administration of any other antitumor therapy
* Have a second primary malignancy that is clinically detectable at the time of consideration for study enrollment
* Have had a prior malignancy other than NSCLC, carcinoma in situ of the cervix, or nonmelanoma skin cancer, unless that prior malignancy was diagnosed and definitively treated at least 5 years previously with no subsequent evidence of recurrence. Patients with a history of low grade (Gleason score ≤6) localized prostate cancer will be eligible even if diagnosed less than 5 years previously
* Patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Difference in terms of quality of life (QOL) between treatment arms | Treatment efficacy will be evaluated at baseline and every 3 cycles during chemo period and every two months during the maintenance phase

SECONDARY OUTCOMES:
treatment activity in terms of response rate | Two year
toxicity evaluation | Two years
Evaluation of QoL across time | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Colucci, MD, Principal Investigator — Oncology Institute of Bari; Domenico Galetta, MD, Study Director — "Giovanni Paolo II" Oncology Instutute Medical Oncology Dept. Bari (Italy)
Locations (12):
- Italy (12):
  - "Giovanni Paolo II" Oncology Institute, Bari, BA
  - "San Paolo Hospital" Oncology Service, Bari, BA
  - Division of Medical Oncology, "Fatebenefratelli" Hospital, Benevento, BN
  - Division of Medical Oncology, "Sen. Perrino" Hospital, Brindisi, Italy, Brindisi, BR
  - 7 Division of Medical Oncology, "Casa Sollievo della Sofferenza" Hospital,, San Giovanni Rotondo, FG
  - Medical Oncology Division "Vito Fazzi" Hospital, Lecce, Le
  - Division of Medical Oncology, "Buccheri-La Ferla" Hospital, Palermo, PA
  - Division of Medical Oncology, "La Maddalena" Hospital, Palermo, PA
  - Division of Medical Oncology, Castellaneta Hospital, Castellaneta, TA
  - Division of Medical Oncology "San Giuseppe Moscati Hospital", Taranto, TA
  - Clinical Trials Office, Department of Medical Sciences, Azienda ULSS 13, Mirano, VE
  - National Cancer Institute "G. Pascale" Thoracic Dept., Napoli

REFERENCES:
- [Derived] Galetta D, Cinieri S, Pisconti S, Gebbia V, Morabito A, Borsellino N, Maiello E, Febbraro A, Catino A, Rizzo P, Montrone M, Misino A, Logroscino A, Rizzi D, Di Maio M, Colucci G. Cisplatin/Pemetrexed Followed by Maintenance Pemetrexed Versus Carboplatin/Paclitaxel/Bevacizumab Followed by Maintenance Bevacizumab in Advanced Nonsquamous Lung Cancer: The GOIM (Gruppo Oncologico Italia Meridionale) ERACLE Phase III Randomized Trial. Clin Lung Cancer. 2015 Jul;16(4):262-73. doi: 10.1016/j.cllc.2014.12.002. Epub 2014 Dec 9. PMID 25582493